CLINICAL TRIAL: NCT04942080
Title: Interest of CALR Allele Burden in Diagnosis and Follow-up of Patients With CALR Mutated Myeloproliferative Syndromes (CALRSUIVI)
Acronym: CALRSUIVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC21_0156
Record Dates: First submitted 2021-06-09; First posted 2021-06-28 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Myeloproliferative Neoplasm; Essential Thrombocythemia; Primary Myelofibrosis, Prefibrotic Stage; Primary Myelofibrosis, Fibrotic Stage
Keywords: CALR; Myeloproliferative Neoplasm; Essential Thrombocythemia; Primary Myelofibrosis; Thrombocytosis
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Primary Myelofibrosis; Thrombocytosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CALRSUIVI cohort (Experimental)
  Interventions: Biological: CALR allele burden quantification

INTERVENTIONS:
Biological: CALR allele burden quantification — * DNA extraction from blood sample for CALR mutation quantification (fragment analysis)
  * at diagnosis and follow-up (inclusion period: 3 years)
  * max 1 sample/year
  * secondary outcome: mutational landscape by Next Generation Sequencing (NGS) analysis at diagnosis

SUMMARY:
Prospective study to evaluate the relevance of CALR allele burden monitoring as a molecular marker of disease progression.

DETAILED DESCRIPTION:
A first local study on 45 patients showed the prognostic impact of CALR mutation quantification in follow-up, independently of the European LeukemiaNet (ELN) prognostic score validated in this group of patients.

This study aims to evaluate a multicenter cohort of 260 patients, including all types of CALR-mutated MPNs and several follow-up samples, to model the temporal evolution of CALR allele burden.

Blood of MPN patients will be collected, at the time of diagnosis and for 3 years (max 1 sample/year), for the quantification of the CALR allele burden. During follow-up, a clinicobiological score to define the progression or not of the disease for each patient will be evaluated in Essential Thrombocythemia (ET) and MyeloFibrosis (MF).

ELIGIBILITY:
Inclusion Criteria:

* adults (age ≥18 years),
* affiliated to the national social security system,
* with CALR mutated myeloproliferative neoplasm diagnosed between 2006 - 2020,
* for which at least one sample is available at the time of diagnosis or before cytoreductive treatment,
* who signed the consent to participate in the study,
* included, or consenting to be included, in the national clinical-biological database of France Intergroupe Syndrome Myéloprolifératifs (FIM).

Exclusion Criteria:

* patient with another active hematological disease or cancer at the time of diagnosis,
* person subject to legal protection scheme or incapable of giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-04-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
For each disease, Hazard Ratio of the different trajectories of CALR allele burden to explain the time to onset of disease progression by the clinicobiological score. | 3 years follow-up
  Clinicobiological score :
  For ET, disease progression if ≥ 1 of:
  * leukocytosis > 12 G/L or myelemia > 10% or erythroblasts > 1%,
  * anemia or thrombocytopenia not related to drug toxicity,
  * development or worsening of splenomegaly,
  * development of thrombocytosis (platelets > 450 G/L) on cytoreductive therapy,
  * poor disease control (at least one change in therapy for reasons other than adverse events),
  * hematologic transformation or death related to hematologic pathology.
  For MF, disease progression if ≥ 1 of:
  * anemia < 100 g/L, neutropenia < 1 G/L, thrombocytopenia < 100 G/L and/or development of general signs not previously present or recurring after improvement,
  * increase in leukocytosis > 25 G/L not previously present,
  * appearance or aggravation of transfusion dependence,
  * appearance (> 5 cm) or aggravation (> 50%) of splenomegaly,
  * leukemic transformation or death related to the hematologic pathology.

SECONDARY OUTCOMES:
A multinomial logistic model will be performed to identify the characteristics associated with the different trajectories of CALR allele burden (pathology, treatment, additional mutations, type of CALR mutation). | 3 years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

REFERENCES:
- [Background] Cottin L, Riou J, Orvain C, Ianotto JC, Boyer F, Renard M, Truchan-Graczyk M, Murati A, Jouanneau-Courville R, Allangba O, Mansier O, Burroni B, Rousselet MC, Quintin-Roue I, Martin A, Sadot-Lebouvier S, Delneste Y, Chretien JM, Hunault-Berger M, Blanchet O, Lippert E, Ugo V, Luque Paz D. Sequential mutational evaluation of CALR -mutated myeloproliferative neoplasms with thrombocytosis reveals an association between CALR allele burden evolution and disease progression. Br J Haematol. 2020 Mar;188(6):935-944. doi: 10.1111/bjh.16276. Epub 2019 Nov 11. PMID 31710700